CLINICAL TRIAL: NCT00005273
Title: Pulmonary Complications of HIV Infection Study (PACS)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1300; U01HL048534 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections; Lung Diseases; Pneumocystis Carinii Infections; AIDS-related Complex
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Lung Diseases; Pneumocystis Infections; AIDS-Related Complex

SUMMARY:
To evaluate the types, incidence, course, and outcome of pulmonary disorders in newly diagnosed cases of Acquired Immune Deficiency Syndrome (AIDS), newly diagnosed cases of AIDS-related complex (ARC) and newly diagnosed asymptomatic human immunodeficiency virus (HIV) infection.

DETAILED DESCRIPTION:
BACKGROUND:

Pulmonary infections as a group are the most commonly recognized life threatening disorders in patients with the AIDS. Although Pneumocystis carinii was the predominant pulmonary pathogen found in these patients, other organisms were clearly of importance as well, not with early years of the HIV epidemic only in patients with AIDS and ARC but in individuals with asymptomatic HIV infection.

In the mid-1980s, physicians who examined many AIDS patients had the impression that a shift was occurring in the types and incidence of pulmonary complications associated with HIV infection. For example, there appeared to be an increased incidence of serious infections caused by pyogenic bacteria and pulmonary and extrapulmonary infection with M. tuberculosis had been noted with increased frequency. Furthermore, lymphoid interstitial pneumonitis (LIP), which is diagnostic of AIDS in children under 13 years old who are HIV antibody positive, was diagnosed with increased frequency in adults. Nonspecific interstitial pneumonitis also appeared to be on the rise. Legionella pneumonia, in contrast to its increased incidence during 1981-83, was now seldom encountered. However, apart from the increased incidence of tuberculosis, a reportable disease, these other shifts in the incidence of pulmonary complications had not been verified.

Because diagnostic strategies in the development of new treatment regimens and new approaches for clinical research were dependent upon knowledge of the incidence and natural history of pulmonary complications associated with HIV infection, the collection of such information was important.

The Request for Proposals for this initiative was released in January 1987. Awards were made in September 1987. The study was funded jointly by the NHLBI and the NIAID. The study was extended by the cooperative agreement mechanism in FY 1993.

DESIGN NARRATIVE:

The cohort consisted of 3 groups: Group A HIV seropositive, no symptoms attributable to HIV and CD4+ Cells >= 400 per microliter; Group B HIV seropositive chemical manifestations of HIV in past 6 months or CD4+ Cells < 400 per microliter; and Group C HIV seronegative controls. The pulmonary status of individuals in each of the categories was evaluated by such methods as chest radiography, pulmonary function tests, nuclear medicine studies, and histological and/or microbiological evaluation. The prospective cohort study described the incidence and course of lung diseases at all stages of HIV infection. Six clinical centers from different geographic areas in the United States began enrolling participants in 1988, and the resulting cohort comprised 1,369 members. HIV seropositive participants were randomized to "intensive" (pulmonary disease screening and follow-up at three-month intervals) or "routine" (six-month follow-up intervals with annual screening) follow-up to assess the impact of these strategies on patient outcomes. The contract-supported phase of the study was jointly funded by the NHLBI and the NIAID.

In 1992, the NHLBI decided to extend follow-up for another five years. The contractors applied for research grants which were approved by the National Heart, Lung, and Blood Advisory Council in May 1992 and awarded in October, 1992. In the renewal, particular attention was given to identifying patterns of complications among demographic subgroups that had not been extensively studied, such as women and Blacks, and to defining differences between HIV transmission groups. The study ended in May, 1997.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1987-09; Study Completion 1997-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Glassroth — Medical College of Pennsylvania; Jeffrey Glassroth — Northwestern University; Philip Hopewell — University of California; Paul Kvale — Henry Ford Hospital; W. Poole — RTI International; Lee Reichman — New Jersey U of Medicine and Dentistry; Lee Reichman — University of Medicine and Dentistry of New Jersey; Mark Rosen — Beth Israel Medical Center; Mark Rosen — Icahn School of Medicine at Mount Sinai; Jeanne Wallace — University of California

REFERENCES:
- [Background] Johnson CC, Wilcosky T, Kvale P, Rosen M, Stansell J, Glassroth J, Reichman L, Wallace J, Markowitz N, Thompson JE, Hopewell P. Cancer incidence among an HIV-infected cohort. Pulmonary Complications of HIV Infection Study Group. Am J Epidemiol. 1997 Sep 15;146(6):470-5. doi: 10.1093/oxfordjournals.aje.a009300. PMID 9290507
- [Background] Chin DP, Osmond D, Page-Shafer K, Glassroth J, Rosen MJ, Reichman LB, Kvale PA, Wallace JM, Poole WK, Hopewell PC. Reliability of anergy skin testing in persons with HIV infection. The pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1982-4. doi: 10.1164/ajrccm.153.6.8665065.
- [Background] Wallace JM, Hansen NI, Lavange L, Glassroth J, Browdy BL, Rosen MJ, Kvale PA, Mangura BT, Reichman LB, Hopewell PC. Respiratory disease trends in the Pulmonary Complications of HIV Infection Study cohort. Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 1997 Jan;155(1):72-80. doi: 10.1164/ajrccm.155.1.9001292.
- [Background] Rosen MJ, Clayton K, Schneider RF, Fulkerson W, Rao AV, Stansell J, Kvale PA, Glassroth J, Reichman LB, Wallace JM, Hopewell PC. Intensive care of patients with HIV infection: utilization, critical illnesses, and outcomes. Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 1997 Jan;155(1):67-71. doi: 10.1164/ajrccm.155.1.9001291.
- [Background] Stansell JD, Osmond DH, Charlebois E, LaVange L, Wallace JM, Alexander BV, Glassroth J, Kvale PA, Rosen MJ, Reichman LB, Turner JR, Hopewell PC. Predictors of Pneumocystis carinii pneumonia in HIV-infected persons. Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 1997 Jan;155(1):60-6. doi: 10.1164/ajrccm.155.1.9001290.
- [Background] Markowitz N, Hansen NI, Hopewell PC, Glassroth J, Kvale PA, Mangura BT, Wilcosky TC, Wallace JM, Rosen MJ, Reichman LB. Incidence of tuberculosis in the United States among HIV-infected persons. The Pulmonary Complications of HIV Infection Study Group. Ann Intern Med. 1997 Jan 15;126(2):123-32. doi: 10.7326/0003-4819-126-2-199701150-00005. PMID 9005746
- [Background] Poole WK, Fulkerson W, Lou Y, Kvale P, Hopewell PC, Hirschtick R, Glassroth J, Rosen M, Mangura B, Wallace J, Markowitz N. Overall and cause-specific mortality in a cohort of homo-/bisexual men, injecting drug users, and female partners of HIV-infected men. Pulmonary Complications of Human Immunodeficiency Virus Infection Study Group. AIDS. 1996 Sep;10(11):1257-64. doi: 10.1097/00002030-199609000-00012. PMID 8883588
- [Background] Schneider RF, Hansen NI, Rosen MJ, Kvale PA, Fulkerson WJ Jr, Goodman P, Meiselman L, Glassroth J, Reichman LB, Wallace JM, Hopewell PC. Lack of usefulness of radiographic screening for pulmonary disease in asymptomatic HIV-infected adults. Pulmonary Complications of HIV Infection Study Group. Arch Intern Med. 1996 Jan 22;156(2):191-5. PMID 8546552
- [Background] Hirschtick RE, Glassroth J, Jordan MC, Wilcosky TC, Wallace JM, Kvale PA, Markowitz N, Rosen MJ, Mangura BT, Hopewell PC. Bacterial pneumonia in persons infected with the human immunodeficiency virus. Pulmonary Complications of HIV Infection Study Group. N Engl J Med. 1995 Sep 28;333(13):845-51. doi: 10.1056/NEJM199509283331305. PMID 7651475
- [Background] Rosen MJ, Lou Y, Kvale PA, Rao AV, Jordan MC, Miller A, Glassroth J, Reichman LB, Wallace JM, Hopewell PC. Pulmonary function tests in HIV-infected patients without AIDS. Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 1995 Aug;152(2):738-45. doi: 10.1164/ajrccm.152.2.7633736.
- [Background] Glassroth J, Jordan M, Wallace JM, Kvale PA, Follmann DA, Rosen MJ, Reichman LB, Mossar M, Hopewell PC. Use of preventive interventions by persons infected with type-1 human immunodeficiency virus (HIV-1). The Pulmonary Complications of HIV Study Group. Am J Prev Med. 1994 Sep-Oct;10(5):259-66. PMID 7848668
- [Background] Kvale PA, Hansen NI, Markowitz N, Rosen MJ, Jordan MC, Meiselman L, Glassroth J, Reichman LB, Wallace JM, Stansell JD, et al. Routine analysis of induced sputum is not an effective strategy for screening persons infected with human immunodeficiency virus for Mycobacterium tuberculosis or Pneumocystis carinii. Pulmonary Complications of HIV Infection Study Group. Clin Infect Dis. 1994 Sep;19(3):410-6. doi: 10.1093/clinids/19.3.410. PMID 7811858
- [Background] Kvale PA, Rosen MJ, Hopewell PC, Markowitz N, Hansen N, Reichman LB, Wallace JM, Glassroth J, Fulkerson W, Meiselman L. A decline in the pulmonary diffusing capacity does not indicate opportunistic lung disease in asymptomatic persons infected with the human immunodeficiency virus. Pulmonary Complications of HIV Infection Study Group. Am Rev Respir Dis. 1993 Aug;148(2):390-5. doi: 10.1164/ajrccm/148.2.390. PMID 8102043
- [Background] Markowitz N, Hansen NI, Wilcosky TC, Hopewell PC, Glassroth J, Kvale PA, Mangura BT, Osmond D, Wallace JM, Rosen MJ, Reichman LB. Tuberculin and anergy testing in HIV-seropositive and HIV-seronegative persons. Pulmonary Complications of HIV Infection Study Group. Ann Intern Med. 1993 Aug 1;119(3):185-93. doi: 10.7326/0003-4819-119-3-199308010-00002. PMID 8100692
- [Background] Wallace JM, Rao AV, Glassroth J, Hansen NI, Rosen MJ, Arakaki C, Kvale PA, Reichman LB, Hopewell PC. Respiratory illness in persons with human immunodeficiency virus infection. The Pulmonary Complications of HIV Infection Study Group. Am Rev Respir Dis. 1993 Dec;148(6 Pt 1):1523-9. doi: 10.1164/ajrccm/148.6_Pt_1.1523. PMID 8256894
- [Background] Design of a prospective study of the pulmonary complications of human immunodeficiency virus infection. The Pulmonary Complications of HIV Infection Study Group. J Clin Epidemiol. 1993 Jun;46(6):497-507. doi: 10.1016/0895-4356(93)90122-h. PMID 8501476
- [Background] Wallace JM, Stone GS, Browdy BL, Tashkin DP, Hopewell PC, Glassroth J, Rosen MJ, Reichman LB, Kvale PA. Nonspecific airway hyperresponsiveness in HIV disease. Pulmonary Complications of HIV Infection Study Group. Chest. 1997 Jan;111(1):121-7. doi: 10.1378/chest.111.1.121. PMID 8996005
- [Background] Osmond DH, Chin DP, Glassroth J, Kvale PA, Wallace JM, Rosen MJ, Reichman LB, Poole WK, Hopewell PC. Impact of bacterial pneumonia and Pneumocystis carinii pneumonia on human immunodeficiency virus disease progression. Pulmonary Complications of HIV Study Group. Clin Infect Dis. 1999 Sep;29(3):536-43. doi: 10.1086/598629. PMID 10530443
- [Background] Huang L, Stansell J, Osmond D, Turner J, Shafer KP, Fulkerson W, Kvale P, Wallace J, Rosen M, Glassroth J, Reichman L, Hopewell P. Performance of an algorithm to detect Pneumocystis carinii pneumonia in symptomatic HIV-infected persons. Pulmonary Complications of HIV Infection Study Group. Chest. 1999 Apr;115(4):1025-32. doi: 10.1378/chest.115.4.1025. PMID 10208204
- [Background] Wallace JM, Lim R, Browdy BL, Hopewell PC, Glassroth J, Rosen MJ, Reichman LB, Kvale PA. Risk factors and outcomes associated with identification of Aspergillus in respiratory specimens from persons with HIV disease. Pulmonary Complications of HIV Infection Study Group. Chest. 1998 Jul;114(1):131-7. doi: 10.1378/chest.114.1.131. PMID 9674459
- [Background] Diaz PT, King MA, Pacht ER, Wewers MD, Gadek JE, Neal D, Nagaraja HN, Drake J, Clanton TL. The pathophysiology of pulmonary diffusion impairment in human immunodeficiency virus infection. Am J Respir Crit Care Med. 1999 Jul;160(1):272-7. doi: 10.1164/ajrccm.160.1.9812089. PMID 10390411
- [Background] Morris AM, Huang L, Bacchetti P, Turner J, Hopewell PC, Wallace JM, Kvale PA, Rosen MJ, Glassroth J, Reichman LB, Stansell JD. Permanent declines in pulmonary function following pneumonia in human immunodeficiency virus-infected persons. The Pulmonary Complications of HIV Infection Study Group. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):612-6. doi: 10.1164/ajrccm.162.2.9912058. PMID 10934095